CLINICAL TRIAL: NCT02968823
Title: Licorice Versus Sugar-water Gargling for Pain in Patients Recovering From Ear-Nose-Throat (ENT) and Maxilla-Facial Surgery - A Randomized, Double-blind Study
Brief Title: Licorice Versus Sugar-water Gargling for Pain in Patients Recovering From Ear-Nose-Throat and Maxilla-Facial Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Olga Plattner, Ao. Univ. Prof., Head of ophthalmologic anesthesia, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1308/2016
Record Dates: First submitted 2016-11-14; First posted 2016-11-21 (Estimated); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Pain, Postoperative; Surgery, Oral
Keywords: Postoperative Pain; Anesthesia; Oral Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Glycyrrhiza glabra extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Licorice (Active Comparator): Licorice gargle
  Interventions: Other: Licorice
- Sugar water (Placebo Comparator): Sugar gargle
  Interventions: Other: Sugar water

INTERVENTIONS:
Other: Licorice — ExtractumLiquiritiaeFluidum, 1 g diluted in 30cc water, gargle the solution for 60 seconds without swallowing it starting preoperatively, 3 times a day until post-operative day 3
  Other Names: Extractum Liquiritiae Fluidum
  Arms: Licorice
Other: Sugar water — Sugar gargle: Sirupus Simplex (sugar 5 g) diluted in 30cc water, gargle the solution for 60 seconds without swallowing it starting preoperatively, 3 times a day until post-operative day 3
  Arms: Sugar water

SUMMARY:
Our primary aim is to determine whether licorice gargling provides meaningful analgesia after oral surgery. Specifically, we propose to test the primary hypothesis that gargling with licorice solution reduces pain after oral surgery more than gargling with sugar water. Because effective analgesia can reduce pain and/or opioid consumption, we will jointly evaluate verbal response pain scores and overall morphine consumption considering licorice to be beneficial only if it proves non-inferior on both measures and superior on at least one.

ELIGIBILITY:
Inclusion Criteria:

1. Oropharyngeal surgeries including:Panendoscopic surgery; elective tonsillectomy/adenotonsillectomy; demarcation and biopsy of suspected tongue carcinoma
2. Anticipated extubation in the operating room
3. American Society of Anesthesia physical status 1-3

Exclusion Criteria:

1. Rapid Sequence Induction
2. Known or suspected allergy to licorice or its ingredients
3. Liver failure with bleeding disorders
4. Insulin-dependent diabetes mellitus
5. Use of non-steroidal anti-inflammatory drug medication within 24 hours before surgery
6. Chronic opioid use
7. Dementia or inability to use an iv Patient-Controlled-Analgesia (PCA) pump
8. superinfected oropharyngeal tumors
9. Planned postoperative mechanical ventilation or admission to Intensive Care Unit (ICU)

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
joint - pain scores and opiate consumption in Post Anesthesia Care Unit (PACU) | first 2 postoperative hours
  A joint outcome of average pain score and total opioid consumption between the end of surgery and the first two postoperative hours. Joint hypothesis testing will be used, meaning that Licorice gargling will be deemed better than sugar-water only if found noninferior on both opioid consumption and pain score and superior on at least one of the two.

SECONDARY OUTCOMES:
joint - pain scores and opiate consumption on day of surgery | from end of surgery until the morning of Post-Operative Day (POD) 1
  Postoperative pain intensity and opioid consumption between the end of surgery and the first postoperative morning. Joint hypothesis testing will be used, meaning that Licorice gargling will be deemed better than sugar-water only if found noninferior on both opioid consumption and pain score and superior on at least one of the two.
joint - pain scores and analgesic consumption | from surgery conclusion to Post-Operative Day (POD) 3
  pain intensity and total analgesics (metamizole or mefenamic acid) consumption in the first three days after surgery. Joint hypothesis testing will be used, meaning that Licorice gargling will be deemed better than sugar-water only if found noninferior on both opioid consumption and pain score and superior on at least one of the two.
postoperative coughing | first 2 postoperative hours
  incidence and intensity of postoperative coughing between surgery and the first two hours in the PACU

CONTACTS AND LOCATIONS:
Overall Officials: Olga Plattner, M.D., Study Chair — Medical University of Vienna; Marita Windpassinger, M.D., Principal Investigator — Medical University Vienna
Locations (1):
- MUVienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No